CLINICAL TRIAL: NCT05227976
Title: Short- and Long-term Effects of Patient Education With or Without Physical Training or Mindfulness and Medical Yoga in Patients With Established Spinal Osteoporosis
Brief Title: Patient Education With or Without Physical Training or Mindfulness and Medical Yoga in Established Spinal Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Anna Spangeus, Associate Professor, MD, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOL-study
Record Dates: First submitted 2022-01-12; First posted 2022-02-08 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Osteoporosis; Vertebral Fracture
Keywords: patient education; yoga; mindfulness; physical training
MeSH Terms: conditions — Osteoporosis; Spinal Fractures | interventions — Patient Education as Topic; Physical Conditioning, Human; Mindfulness; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Theory only (Active Comparator): Once weekly for 10 weeks
  Interventions: Behavioral: Patient education (Theory)
- Theory and physical training (Active Comparator): Once weekly for 10 weeks
  Interventions: Behavioral: Patient education (Theory); Behavioral: Physical training
- Theory and mindfulness/medical yoga (Active Comparator): Once weekly for 10 weeks
  Interventions: Behavioral: Patient education (Theory); Behavioral: Mindfulness and medical yoga in group

INTERVENTIONS:
Behavioral: Patient education (Theory) — Theory/Lectures (1h/week)
  Interventions given once weekly for 10 weeks.
Behavioral: Physical training — Physical training group (1 hour/week)
  Interventions given once weekly for 10 weeks.
  Arms: Theory and physical training
Behavioral: Mindfulness and medical yoga in group — Mindfulness/medical yoga in group (1hour/week)
  Interventions given once weekly for 10 weeks.
  Arms: Theory and mindfulness/medical yoga

SUMMARY:
In the present feasibility and pilot study we aim to investigate the effect and safety of patient education with or without additional physical training or mindfulness/medical yoga in patients with manifest spinal osteoporosis (at least one vertebral fracture).

The study includes a 10-week intervention period with once weekly theory education with or without additional physical training or mindfulness/medical yoga (randomized groups). Furthermore, a proceeding observation period of 10 weeks as well as a 1-year follow up post-intervention observation are included in the study design.

DETAILED DESCRIPTION:
The SOL-study (School of Osteoporosis in Linköping) is a feasibility and pilot study on patient education in manifest spinal osteoporosis. The study design is interventional with patients randomized to one of three different interventions, i.e.

1. Theory only (T group)
2. Theory and physical exercise (TPh-group)
3. Theory and mindfulness/medical yoga (TMMY-group)

The intervention period is 10 weeks, including 1 hour theory session/week (same for all groups) and for TPh- and TMMY-groups a one hour group training session is scheduled before the theory session.

Inclusion criteria are: 1) manifest spinal osteoporosis (diagnosed osteoporosis and > 1 vertebral fracture [VF]); 2) > 3 months had passed since the most recent VF; and 3) age over 60 years.

Clinical testing and questionnaire evaluation are performed at three timepoints; 1) Baseline (T1), i.e. before intervention; 2) Post-observation (T2) i.e. after a passive observation time of 4 months); and 3) Post-intervention (T3) i.e. after the interventions. A one year follow up post-intervention is performed by questionnaire evaluation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with established spinal osteoporosis (at least one vertebral fracture and osteoporosis)
* >3 months had passed since the most recent VF
* age ≥60 years
* physical ability to walk without an indoor walker

Exclusion Criteria:

* inability to understand the Swedish language or difficulty following the research protocol or dementia

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (HRQoL) - disease specific | 1.5 year
  Assessed with Qualeffo-41 (quality of life questionnaire of the European foundation for osteoporosis). The Qualeffo-41 includes 41 questions in seven domains. Domain scores are calculated by averaging the scores of one domain, and transforming them into a 0-100 scale according to a manual on scoring algorithm. Zero indicates the best possible and 100 the worst HRQoL. The Total Qualeffo-41 score is calculated by summing the answers of all questions and transforming the raw total scores from 0-100 (IOF homepage 2007 http://www.iofbonehealth.org)
Health-related quality of life (HRQoL) - generic | 1.5 year
  Assessed with RAND-36 (Research and Development questionnaire). The RAND-36 compromises 36 items with two to six response options according to an ordinal scale. Eight health domains are assessed, coded, scored and summarised to derive the domains. The scores are transformed into a 0-100 scale. Zero indicates the worst possible HRQoL and 100 the best.
Body weight | 6 months
  Body weight (kg) is measured by a digital scale, and with the participant in an upright position without shoes.
Body height | 6 months
  Body height (cm) is measured by a stadiometer with the participant in an upright position without shoes.
Static balance test | 6 months
  The static balance tests are performed without shoes both with the eyes open and with the eyes closed. (The floor is leveled, and the room is well illuminated). The static balance tests are limited to a maximum of 30 seconds and timed by using a stop-watch. The one-leg stance tests are performed with the opposite foot lifted halfway upon the calf of the supported leg and the arms at a vertical position at the sides of the body. If the participant has contact with the floor with the non-standing foot the time is stopped. The one-leg standing time (on each leg) tests are performed three times and the best of the trials is used as the final score
Dynamic balance test | 6 months
  Dynamic balance tests are walking without shoes forwards heel to toe on a line and walking backwards toe to heel on a line. These tests are performed three times and the number of correct steps is counted and maximized to 15 correct steps, where the best of the trials is used as the final score.
Muscle strength Chair-stand | 6 months
  The chair-stand test is performed from sitting on a stable chair with the arms crossed in front of the chest. The total number of risings is counted for 30 seconds using a stop-watch.
Muscle strength Hand grip | 6 months
  Hand grip strength is measured in kilograms by using the Jamar dynamometer both of the dominant and the non-dominant hand. The subject is sitting on a stable chair with 90° of the elbow and support for the forearm in a neutral position, but with no support for the hand which is gripping the dynamometer. The adjustable handle was set at the second handle position for standardization. Each test was performed three times and the best trial was used as the final score.
C7 to wall distance | 6 months
  The participant stans upright, as tall as possible, with both heels and the back against the wall and the head in a neutral position. A folding ruler is used to measure the perpendicular distance in centimeter between the seventh cervical vertebra (C7) and the wall.
Pain assessment | 1.5 year
  Numeric rating scale (NRS) is used to measure present pain intensity, pain for the last week and worst pain. The participant is asked to report an integer between 0-10 to assess the perceived pain, where "no pain" is rated as 0 and "worst possible pain" is rated as 10.
Number of patients using pain medications regularly | 1.5 year
  Participants are asked for their usage of pain medications (i.e. names of the drugs).
Physical activity | 1.5 year
  Two physical activity questions are used and answered by categories on a six-point (question 1) and seven-point Likert scale (question 2), respectively:
  1. First question: During a regular week, how much time do you spend exercising on a level that makes you short winded, for example running, fitness class or ball games? Possible answers: 0 minutes, <30 minutes, 30-60 minutes, 60-90 minutes, 90-120 minutes, >120 minutes (
  2. Second question: During a regular week, how much time are you physically active in ways that are not exercise, for example walks, bicycling or gardening? Add together all activities lasting at least 10 minutes. Possible answers: 0 minutes, <30 minutes, 30-60 minutes, 60-90 minutes, 90-150 minutes, 150-300 minutes, >300 minutes
Patient enablement instrument (PEI) | 1.5 year
  The patient enablement instrument (PEI) is used to measure the patient's perceived change in ability to understand and cope with his or her health issues after the treatment period and contains six items. The text "As a result of the participating in the Osteoporosis School, do you feel that you are …" is followed by six items; 1) able to cope with life, 2) able to understand your illness, 3) able to cope with your illness, 4) able to keep yourself healthy, 5) confident about your health, and 6) able to help yourself. The following five alternative answers were used for each statement; much better/much more, better/more, same, less/worse and not applicable. The PEI point for much better/much more is 2; for better/more is 1; and for same, less/worse or not applicable is 0. These points are added and thus the total PEI score ranges between 0 (worst score) and 12 (best score).
Subjective experience of the patient education | 1.5 year
  The participants' overall experiences of the theoretical lectures (and the physical training) are scored on a six-level Likert scale (scores 0-6), where 5 is considered very satisfied and 0 is not at all satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Spångeus, Ass.Prof, MD, Principal Investigator — Univerity Hospital Linköping, Linköping University
Locations (1):
- University Hospital Linköping, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No